CLINICAL TRIAL: NCT01224418
Title: Clinical Study to Evaluate the Efficacy of Tacrolimus in Active Rheumatoid Arthritis Patients Shown Unsuccessful Response Against Methotrexate: Non-comparative, Single Arm, Multi-center, Phase 4 Study
Brief Title: A Study to Evaluate the Efficacy of Tacrolimus in Rheumatoid Arthritis Patients Shown Unsuccessful Response to Methotrexate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRGRA-08-01-KOR
Record Dates: First submitted 2010-10-14; First posted 2010-10-20 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Tacrolimus; Prograf; Calcinurin inhibitor; Rheumatoid arthritis(RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus group (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — oral
  Other Names: Prograf; FK506

SUMMARY:
This study is to evaluate efficacy of 6 months treatment of tacrolimus in active Rheumatoid Arthritis patients who showed unsuccessful response against methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with more than 6 months history of rheumatoid arthritis according to ACR criteria
* Patients who have been treated unsuccessfully to more than single DMARDs including methotrexate at the discretion of investigator
* ESR ≥ 30 mm/h or CRP ≥ 1.0 mg/dL (ESR: Erythrocyte Sedimentation Rate, CRP: C-Reactive Protein)
* Patients are required to have at least 3 of 66 joints assessed as swollen
* Patients are required to have at least 6 of 68 joints assessed as painful with pressure

Exclusion Criteria:

* Pregnant or breast-feeding patients. Patients who plan to bear children or breast-feed during the study and within 6 month after completion of study
* Previous experience of tacrolimus (ointment excluded)
* Renal impairment or serum creatinine > 1.4 mg/dL
* Liver function failure as follows: viral hepatitis, non-viral hepatitis, cirrhosis, SGOT/SGPT > 2x upper limit normal
* Patients with history of pancreatitis, glucose intolerance or complication or who indicates any of the following criteria:Blood glucose level >110mg/dl before the meal and >200mg/dl after the meal HbA1c > 6.4%
* Cardiac disease(ischemic heart disease, treatment-requiring arrhythmia, heart failure)or complications
* Other investigational drug within last 30 days
* Patients who have been treated with infliximab, adalimumab, or leflunomide within 8 weeks of start of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
ACR20 response rate compared to baseline | Baseline and up to 6 months
  (ACR20: 20% improvement in American College of Rheumatology Core Set)

SECONDARY OUTCOMES:
ACR50 response rate compared to baseline | Baseline and up to 6 months
ACR70 response rate compared to baseline | Baseline and up to 6 months
Changes from baseline in 100mm pain VAS (Visual Analogue Scale) | Baseline and up to 6 months
Safety assessed by the incidence of adverse event and abnormalities in clinical laboratory test | For 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (2):
- South Korea (2):
  - Gyeonggido
  - Seoul